CLINICAL TRIAL: NCT02048761
Title: Locally Delivered 1% Metformin Gel in the Treatment of Intrabony Defects in Subjects With Chronic Periodontitis : A Randomized Controlled Clinical Trial
Brief Title: Locally Delivered 1% Metformin Gel in the Treatment of Intrabony Defects in Chronic Periodontitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2013-14/B
Record Dates: First submitted 2014-01-23; First posted 2014-01-29 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Intrabony Defects in Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo Group (Placebo Comparator): After debridement, placebo gel was applied into the periodontal pockets with a syringe and a blunt canula.
  Interventions: Drug: Placebo gel
- 1% Metformin (Active Comparator): After debridement, 1% Metformin gel was applied into the periodontal pockets with a syringe and a blunt canula.
  Interventions: Drug: 1 % Metformin gel

INTERVENTIONS:
Drug: Placebo gel — After debridement, a single dose of the placebo gel was applied into the periodontal pockets with a syringe and a blunt canula
  Arms: Placebo Group
Drug: 1 % Metformin gel — After debridement, 1% Metformin gel gel was applied into the periodontal pockets with a syringe and a blunt canula.
  Arms: 1% Metformin

SUMMARY:
This study was designed as a randomized, controlled clinical trial to evaluate the efficacy of 1% MF gel as local drug delivery in adjunct to SRP for the treatment of intrabony defects in chronic periodontitis in comparison with placebo gel.

DETAILED DESCRIPTION:
Background: Metformin (MF) belonging to the class biguanide, is a first-line therapy for type 2 diabetes mellitus, and is one of the most commonly prescribed oral hypoglycemic drug worldwide. MF has shown to posses bone forming and bone sparring actions. The present study was designed to investigate effectiveness of MF, 1 % in an indigenously prepared biodegradable controlled-release gel as, as an adjunct to scaling and root planing (SRP) in treatment of chronic periodontitis subjects with intrabony defects.

Materials and Methods: Sixty five subjects were categorized into two treatment groups: SRP plus 1% MF and SRP plus placebo. Clinical parameters were recorded at baseline and at 3 and 6 months; they included plaque index (PI), modified sulcus bleeding index (mSBI), probing depth (PD), and clinical attachment level (CAL). At baseline and after 6 months, radiologic assessment of intrabony defect (IBD) fill was done using computer-aided software.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy subjects
* Sites with probing depth (PD) ≥5 mm
* Clinical attachment level (CAL) ≥4 mm
* Vertical bone loss ≥3 mm on intraoral periapical radiographs with no history of periodontal therapy or use of antibiotics in the preceding 6 months were included

Exclusion Criteria:

* Patients with known systemic disease
* Known or suspected allergy to the MF/ biguanide group
* Patients on systemic MF or other oral antidiabetic therapy
* Patients with aggressive periodontitis
* Patients with diabetes
* Use of tobacco in any form
* Alcoholism
* Immunocompromised patients
* Pregnant or lactating females

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Defect depth reduction | Baseline to 6 months
  The primary outcome of the study is to determine the defect depth reduction by 1% metformin gel radio-graphically and compare the outcome with control group.

SECONDARY OUTCOMES:
Probing depth | Baseline to 6 months
  Probing depth is measured from baseline to 3 months and 6 months in both control and test group.
Clinical attachment level | Baseline to 6 months
  Clinical attachment level is measured from baseline to 3 months and 6 months in both control and test group.
Modified sulcular bleeding index | Baseline to 6 months
  Modified sulcular bleeding index is measured from baseline to 3 months and 6 months in both control and test group.
Plaque index | Baseline to 6 months
  Full mouth and site specific plaque index is measured from baseline to 3 months and 6 months in both control and test group.

CONTACTS AND LOCATIONS:
Overall Officials: A R Pradeep, M.D.S., Principal Investigator — Govt Dental College & Research Inst, Bangalore.
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India